CLINICAL TRIAL: NCT06620562
Title: Improving Efficacity of Sleeve Gastrectomy With Naltrexone/Bupropion Extended-release Tablet - A Randomized Controlled Trial
Brief Title: Improving Efficacity of Sleeve Gastrectomy With Naltrexone/Bupropion Extended-release Tablet
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Bausch Health Canada (Unknown)
Responsible Party: Principal Investigator, Laurent Biertho, Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sleeve-Plus
Record Dates: First submitted 2024-08-06; First posted 2024-10-01 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Drug; Obesity, Morbid
MeSH Terms: conditions — Obesity; Obesity, Morbid | interventions — Naltrexone; Bupropion

STUDY DESIGN:
Intervention Model Description: This is a single-center double-blind randomized placebo-controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naltrexone/Bupropion (Experimental): Patients will be started one month after sleeve gastrectomie on a progressive dose of Naltrexone/Bupropion extended-release 8mg/90mg, up to 2 tabs twice a day (32mg/360mg) adjusted according to tolerance and side-effects.
  Interventions: Drug: Naltrexone/Bupropion
- Placebo (Placebo Comparator): Patients will be started one month after sleeve gastrectomie on a progressive numbers of matched placebo tablets up to 2 tabs twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone/Bupropion — Patient randomized in the Neltrexone/Bupropion group will be started one month after surgery on a progressive dose of Naltrexone/Bupropion extended-release 8mg/90mg, up to 2 tabs twice a day (32mg/360mg) adjusted according to tolerance and side-effects to improve long-term use. Duration of therapy will be 24 months.
  Arms: Naltrexone/Bupropion
Drug: Placebo — Patient randomized in the placebo group will be started one month after surgery on a progressive numbers of matched placebo tablets up to 2 tabs twice a day. Duration of therapy will be 24 months.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess the impact of combination therapy with Naltrexone-Bupropion (NB) in the post-operative period of sleeve gastrectomy (SG). on a) weight loss, b) resolution of comorbidities and c) eating behaviors.

Researchers will compare SG-NB group with SG-placebo group to see if they experience significantly higher excess weight loss (EWL) at 12 and 24 months and if there is a significantly higher percentage of patients with an EWL above 50% in the SG-NB group versus in the SG-placebo group.

Participants will be randomized 1:1 to SG in combination with NB versus SG with placebo. Patients will be started one month after surgery on a progressive dose of Naltrexone/Bupropion extended-release or placebo. Duration of therapy will be 24 months.Both groups will benefit from behavioral and nutritional support.

ELIGIBILITY:
Inclusion Criteria:

* MBI above 30 kg/m2 with obesity-related comorbidity or above 35 kg/m2 without associated comorbidities.

Exclusion Criteria:

* Revisional or reoperative surgery
* Pregnancy or planned pregnancy in the next 24 months
* Simultaneous use of other weight loss medication
* Uncontrolled hypertension
* Chronic opioid use or opiate agonist (e.g., methadone) or partial agonists (e.g., buprenorphine) use, or acute opiate withdrawal.
* Use of other bupropion-containing products
* Concomitant administration of monoamine oxidase inhibitors.
* End-stage liver or kidney disease
* Concomitant use of CYP2B6 inhibitors (ticlopidine or clopidogrel)
* Concomitant administration of the antipsychotic thioridazine
* Seizure disorder or a history of seizures
* Cardiac pacemaker
* Current or prior diagnosis of bulimia or anorexia nervosa

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Weight loss | baseline to 24 months
  % Excess weight loss
Percentage of participant with an Excess Weight Loss above 50% | Baseline to 24 months

SECONDARY OUTCOMES:
Resolution of associated comorbidities | Baseline to 24 months
  Type 2 diabetes, hypertension and dislipidemia
Improvement of Eating behaviors (Food Craving State Questionnaire) | Baseline to 24 months
  Evaluates severity of cravings using a validated questionnaire. Minimum : 15; Maximum : 75; Higher scores mean a worse outcome.
Improvement of Eating behaviors (Food Craving Trait Questionnaire) | Baseline to 24 months
  Evaluates severity of cravings using a validated questionnaire. Minimum : 39; Maximum : 234; Higher scores mean a worse outcome.
Decrease in food explicit and implicit wanting and liking food reward. | Baseline to 24 month
  Decrease in food explicit and implicit wanting and liking food reward assessed by Leeds Food Preference Questionnaire using a computerized behavioural task
Improvement in well-being, mood and Quality of Life (SF-36) | Baseline to 24 months
  36-item short form survey evaluating quality of life on a scale from 0 to 100, higher scores indicate better quality of life
Improvement in well-being, mood and Quality of Life (QLaval) | Baseline to 24 months
  Laval questionnaire evaluating quality of life on 6 aspects on a scale from 0 to 7, higher scores indicate better quality of life
Improvement in well-being, mood and Quality of Life (HAD questionnaire) | Baseline to 24 months
  HAD questionnaire includes 14 rated items from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), obtaining two scores (maximum score of each score = 21). Higher scores indicate a worse outcome
Gastro-intestinal side-effects | Baseline to 24-month
  Gastro-intestinal side-effects assessed by GIQLI questionnaire on a scale from 0 to 144. Higher scores indicate better quality of life
Improvement of Eating behaviors (Binge Eating Scale) | Baseline to 24 months
  To assess the presence of certain binge eating behaviors that may be indicative of an eating disorder.
  The higher the score, the more binge eating behaviors is observed. The minimum score is 0 while the maximum score is 46. The final result allows to say if the person has an absent (less than 17), moderate (between 18 and 26) or severe (more than 27) binging level.
Improvement of Eating behaviors (YFAS 2.0) | Baseline to 24 months
  The YFAS 2.0 was designed to assess food addiction. It assesses the symptoms of food addiction and the resulting distress and impaired functioning.
  The higher the level of symptoms, the more severe the food addiction. Impaired functioning and distress are scored from 0 to 2. Symptoms are scored from 0 to 11. If the functioning and distress score is 1 and above, the food addiction may be mild (2-3 symptoms), moderate (4-5 symptoms), or severe (6+ symptoms).

CONTACTS AND LOCATIONS:
Locations (1):
- Criucpq-Ul, Québec, Quebec, Canada